CLINICAL TRIAL: NCT06082700
Title: Correlation Between Missing Posterior Teeth and Vertical Dimension Cephalometric Measurements With Temporomandibular Disorders in a Sample of Adult Egyptian Subjects: A Cross-Sectional Study
Brief Title: Correlation Between Missing Posterior Teeth and Vertical Dimension Measurements With Temporomandibular Joint Disorders in a Sample of Adult Egyptian Subjects
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amir Karam Fahmy Agaiby, master's degree student, Cairo University
Other Study IDs: 13 5 23
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Correlation Between Missing Posterior Teeth and Vertical Dimension Cephalometric Measurements With Temporomandibular Disorders
MeSH Terms: interventions — Diagnostic Imaging; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Diagnostic Test: imaging — clinical examination to see missing posterior teeth & vertical measurements by lateral cephalometric x-ray
  Other Names: clinical examination

SUMMARY:
The goal of this observational study is to learn about the correlation between missing posterior teeth and vertical dimension cephalometric measurements with temporomandibular disorders in a sample of adult Egyptian subjects in. The main questions it aims to answer are:

* Is there a correlation between missing posterior teeth and temporomandibular disorders?
* Is there a correlation between vertical dimension cephalometric measurements and temporomandibular disorders? Participants will be asked for the following:-

  * to give their phone numbers & it will be collected through the orthodontic department patient's database ensuring complete confidentiality.
  * to fill Personal data chart (name, age, date of birth, mobile number, address).
  * to receive Clinical examination to determine number of missing teeth.
  * to receive Clinical examination to diagnose TMD using the DC/TMD.
  * to do Lateral cephalometric radiograph to measure the vertical dimension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with 2 or more missing posterior teeth seeking treatment at the faculty.
* Age: 16-49 years.

Exclusion Criteria:

* - Patients who refuse to participate in the study.
* Patients younger than 16 years.
* Subjects who received previous TMD treatment.
* Subjects suffering from systemic conditions which may affect the functioning of TMJ, for example, rheumatoid arthritis, scleroderma, and septic arthritis.
* Subjects with a history of trauma to the maxillofacial area.
* Subjects with a previous history of maxillofacial surgery.
* Subjects with a history of malignancy or current malignancy of the maxillofacial area.

Ages: 16 Years to 49 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adult Male and female patients with 2 or more missing posterior teeth seeking treatment at the faculty. Age: 16-49 years.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
temporomandibular disorder | 3 months
  will see the Correlation Between Missing Posterior Teeth and Vertical Dimension cephalometric measurements with Temporomandibular Disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No